CLINICAL TRIAL: NCT06354634
Title: Clinical and Radiographic Success of Resin Polymer (NuSmile BioFlx) Compared to Stainless Steel (3M ESPE) Crowns for Restoration of Primary Molar Teeth: a Split Mouth Randomized Controlled Trial.
Brief Title: Resin Polymer (NuSmile BioFlx) Compared to Stainless Steel Crowns (3M ESPE) for Restoration of Primary Molar Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM20028439
Record Dates: First submitted 2024-03-27; First posted 2024-04-09 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Dental Caries; Tooth Decay
MeSH Terms: conditions — Dental Caries | interventions — Crowns

STUDY DESIGN:
Intervention Model Description: Each participant will receive both interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All participants (Experimental): Each participant will receive a BioFLX crown and a stainless steel crown.
  Interventions: Other: Resin polymer (NuSmile Bioflx) crown; Other: Stainless steel crown

INTERVENTIONS:
Other: Resin polymer (NuSmile Bioflx) crown — Resin polymer (NuSmile Bioflx)crown
Other: Stainless steel crown — Stainless steel crown

SUMMARY:
The purpose of this research study is to test the effectiveness of two different crowns/caps on teeth for restoration of primary molar teeth. The two different materials of crowns are resin polymer and stainless steel crowns. These crowns are placed on the teeth to restore function and prevent further caries and infection.

DETAILED DESCRIPTION:
There is a lack of literary evidence for assessment of the properties of Bioflx crowns and their effect on clinical outcomes and parental satisfaction compared to traditionally available options including stainless steel crowns and zirconia crowns. Hence, this study plans to assess the clinical performance and child and parental satisfaction of Bioflx compared to the "gold standard" stainless steel crowns in pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Age: Children age group 3-7 yrs old
* Primary molars affected with caries or hypoplastic defect.
* Occlusion: Primary molar must have antagonist tooth.
* Consent of parent (legal guardians) and child assent for 7 years.
* Multi-surface dental caries observed in more than one tooth, in either side of the same arch (maxilla or mandible) or opposite arch (maxilla or mandible)
* Status: Asymptomatic or symptomatic teeth with signs of reversible pulpitis

Exclusion Criteria:

* Teeth with advanced stages of resorption (more than 2/3rd)
* Teeth exhibiting irreversible pulpitis.
* Teeth for which pulpotomy is done.
* Molar in infraocclusion
* Medically compromised children (ASA 3 or 4)
* History of grinding or pathological attrition
* Adverse gingival or periodontal conditions

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2024-06-07 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
The success of Bioflx crown in primary molars in comparisons with stainless steel molars through clinical assessments | 3, 6, 12, 18, 24 and 36 months
  The clinical outcomes will be measured and reported in the data table based on the number of participants scored on 3-point Likert scale (Ideal, Acceptable, or Not Acceptable) for the following parameters separately: Contour of crown, gingival health, staining of crown, surface roughness of crown, opposing tooth, color match of crown, marginal fit, marginal discoloration, recurrent caries.
The success of Bioflx crown in primary molars in comparisons with stainless steel molars through radiographic assessments | 3, 6, 12, 18, 24 and 36 months
  The radiographic outcomes will be measured and reported in the data table based on the number of participants scored on either presence or absence (yes / no) of the findings for the following parameter separately: Widening of periodontal ligament space, furcation radiolucency, periapical pathology, alveolar crestal bone loss, internal root resorption and external root resorption.

SECONDARY OUTCOMES:
Parental satisfaction | 3, 12, 24 and 36 months
  The questionnaire is a Likert scale of 1-5. 1 equals very dissatisfied. 5 equals very satisfied. The higher the score, the better.
Child satisfaction | 3, 12, 24 and 36 months
  The questionnaire is a Likert scale of 1-5. 1 equals very dissatisfied. 5 equals very satisfied. The higher the score, the better.
ECOHIS (Early Childhood Oral Health Impact Scale) survey | Pre-operative, 6, 12, 24 and 36 months
  The questionnaire is a Likert scale of 1-5. 1 equals never. 5 equals very often. The lower the score, the better.

CONTACTS AND LOCATIONS:
Overall Officials: Jayakumar Jayaraman, BDS, MDS, FDSRCS, MS, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No